CLINICAL TRIAL: NCT07321795
Title: Osteoporotic Vertebral Compression Fractures: A Multi-center Cohort Study Based on Disease and Syndrome Differentiation
Brief Title: Osteoporotic Vertebral Compression Fracture Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other); Suzhou TCM Hospital Affiliated to Nanjing University of Chinese Medicine (Unknown); Shandong Wendeng Orthopedic Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: WJEC-KT-2025-047-P001
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: OVCF Database; Cohort Study
Keywords: Osteoporotic Vertebral Compression Fractures; Traditional Chinese Medicine; Potential biomarkers; Risk prediction model

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human biological samples include serum and plasma. Serum is obtained by allowing whole blood to clot and then centrifuging to remove cells and clotting factors.
  Plasma is obtained by centrifuging anticoagulated whole blood, retaining clotting factors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal bone mass group
- osteopenia group
- osteoporosis group
- Osteoporotic Vertebral Compression Fracture group

SUMMARY:
The study aims to construct an early warning model for Osteoporotic Vertebral Compression Fracture (OVCF) by integrating TCM syndrome patterns with modern risk factors. This is a multi-center cohort study on OVCF integrated with disease and syndrome differentiation in Traditional Chinese Medicine (TCM).

DETAILED DESCRIPTION:
The subjects are selected according to the inclusion criteria and exclusion criteria. A total of 200 subjects will be recruited from four participating tertiary hospitals and categorized into four groups: individuals with normal bone mass, osteopenia, osteoporosis, and Osteoporotic Vertebral Compression Fracture (OVCF) . Data collection encompasses three levels:

* Macro-level: Demographics, lifestyle, medical history, and physical metrics.
* Meso-level: TCM syndrome diagnoses, bone mineral density (BMD), MRI assessments, and functional scores (VAS, ODI).
* Micro-level: Serum biomarkers related to bone metabolism, lipids, inflammation, and muscle health.

Strict quality control measures will be implemented, including researcher training and data monitoring. The integrated database and analytical framework are designed to develop a practical, population-specific risk prediction tool for OVCF.

ELIGIBILITY:
Inclusion Criteria:

1.50 years ≤ age < 80 years; gender includes both male and female. 2.Meet the diagnostic criteria for new-onset osteoporotic vertebral compression fracture.

3.Voluntarily participate in this clinical study and sign the informed consent form.

Subjects meeting only criteria (1) and (3) with a T-score ≥ -1.0 can be included in the normal bone mass group. Subjects meeting criteria (1) and (3) with -2.5 < T-score < -1.0 can be included in the osteopenia group. Subjects meeting criteria (1) and (3) with T-score ≤ -2.5, meeting the diagnostic criteria for osteoporosis, can be included in the OP group. Subjects meeting all criteria (1), (2), and (3) will be included in the OVCF patient group.

Exclusion Criteria:

1. Patients with serious concomitant cardiovascular/cerebrovascular diseases, liver/kidney diseases, malignant tumors, or other wasting diseases, and patients with infectious diseases.
2. Patients with other endocrine system diseases, such as Cushing's syndrome, hyperthyroidism, hypothyroidism, etc.
3. Patients who have participated in other clinical trials within the past 3 months.
4. Patients with concomitant Alzheimer's disease, mental illnesses or depression, or those unable to cooperate to complete the trial.
5. Patients with poor compliance

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants are selected from patients admitted to four participating tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | Baseline
  DXA will be used to measure lumbar spine (L1-L4) and bilateral hip density, recording the T-score for each site. Instrument precision will be set to 1% (i.e., repeated measurement error < 1%). Professionals will be responsible for post-use accuracy checks and maintenance.

SECONDARY OUTCOMES:
Muscle Strength | Baseline
  Left and right handgrip strength in kilograms, which is determined by a handheld dynamometer. The normal range varies by age, gender, and dominant hand. When it is lower than the normal range, it may indicate muscle weakness, sarcopenia, or neuromuscular disorders; when it is higher than the normal range, it typically reflects good musculoskeletal health and physical fitness.
The bone marrow fat fraction (FF) | Baseline
  The bone marrow fat fraction (FF) of lumbar vertebrae (expressed as a percentage), which is determined by magnetic resonance imaging (MRI) analysis. The normal range varies with age and vertebral level, typically between 30-50% in healthy adults. When it is higher than the normal range, it may indicate osteoporosis, aging, or metabolic bone disease; when it is lower than the normal range, it may suggest conditions such as bone marrow edema, inflammation, or hematopoietic disorders.
Paravertebral muscle area | Baseline
  The paravertebral muscle area (in cm²), which is determined by magnetic resonance imaging (MRI) analysis. The normal range varies based on vertebral level, age, and gender. When it is smaller than the normal range, it may indicate muscle atrophy, sarcopenia, or degenerative changes.
Fatty infiltration | Baseline
  The degree of paravertebral muscle fatty infiltration (expressed as a percentage or fat fraction), which is determined by magnetic resonance imaging (MRI) analysis. The normal range varies with age and vertebral level. When it is higher than the normal range, it indicates increased intramuscular fat deposition, often associated with aging, disuse, or metabolic disorders.
Vertebral bone quality (VBQ) score | Baseline
  The vertebral bone quality (VBQ) score, which is determined by magnetic resonance imaging (MRI) analysis. The normal range is 1.5-3.0. When it is higher than the normal range, it indicates poor bone quality and an increased risk of osteoporotic vertebral fractures; when it is lower than the normal range, it indicates better bone quality and a lower fracture risk.
Visual Analogue Scale (VAS) Score | Baseline
  Draw a straight line with a length of 10 cm on the white paper and mark "painless" and "severe pain" on both ends respectively to form VAS. The patient makes a mark on the straight line according to the degree of pain he feels. The distance from the starting point to the mark is the quantified degree of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. Draw a 10 cm long on a piece of white paper.
Lumbar Oswestry Disability Index (ODI) Score | Baseline
  The ODI is a patient-reported questionnaire consisting of 10 sections (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). Each section is scored from 0 to 5, with higher scores indicating greater disability. Interpretation of ODI Scores:0-20%: Minimal disability (can perform daily activities normally).21-40%: Moderate disability (pain and functional limitations affect some activities).41-60%: Severe disability (pain significantly restricts daily life).61-80%: Crippling disability (most activities are severely limited).81-100%: Bed-bound or exaggerated symptoms.
OP TCM Syndrome Information | Baseline
  Four patterns including Kidney Yang Deficiency, Spleen-Kidney Yang Deficiency, Liver-Kidney Yin Deficiency, Kidney Deficiency with Blood Stasis. Two professional TCM clinicians will independently determine the patient's syndrome pattern. In case of disagreement, a third physician will adjudicate.
OVCF TCM Syndrome Information | Baseline
  Four patterns including Qi Stagnation and Blood Stasis, Kidney Deficiency with Blood Stasis, Liver-Kidney Yin Deficiency. Two professional TCM clinicians will independently determine the patient's syndrome pattern. In case of disagreement, a third physician will adjudicate.
Total Type I Procollagen N-terminal Propeptide (P1NP)、β-Cross-linked C-telopeptide of Type I Collagen (β-CTX) | Baseline
  Serum level of Beta-CrossLaps (β-CTX) in ng/mL, N-terminal propeptide of type l procollagen (P1NP) in ng/mL, which are determined by Electrochemiluminescence Method.The normal reference ranges of serum P1NP and ß-CTX are 16.3-78.2 ng/mL and 0.114-0.628 ng/mL, respectively.In case of abnormal conditions,the higher the β-CTX,the more serious the bone resorption.The lower the P1NP, the less bone formation and the worse the bone condition.
Serum bone glaprotein (BGP) | Baseline
  Serum level of bone glaprotein (BGP) in ug/L, which is determined by automatic biochemical analysis The normal value 48-10.2 ug/L.When it is lower than the normal value, it indicates that bone formation is reduced.
25-Hydroxyvitamin D (25(OH)D) | Baseline
  Serum level of 25-Hydroxyvitamin D (25(OH)D) in nmol/L, which is determined by automatic biochemical analysis. The normal value is 50-125 nmol/L. When it is lower than the normal value, it indicates vitamin D deficiency or insufficiency.
Intact Parathyroid Hormone (PTH) | Baseline
  Serum level of Intact Parathyroid Hormone (PTH) in pg/mL, which is determined by automatic biochemical analysis. The normal value is 15-65 pg/mL. When it is higher than the normal value, it may indicate hyperparathyroidism; when it is lower than the normal value, it may indicate hypoparathyroidism or vitamin D intoxication.
Total Cholesterol (TC) | Baseline
  Serum level of Total Cholesterol (TC) in mmol/L, which is determined by automatic biochemical analysis. The normal value is <5.2 mmol/L. When it is higher than the normal value, it indicates an increased risk of cardiovascular disease; when it is lower than the normal value, it may be associated with malnutrition or liver dysfunction.
Triglycerides (TG) | Baseline
  Serum level of Triglycerides (TG) in mmol/L, which is determined by automatic biochemical analysis. The normal value is <1.7 mmol/L. When it is higher than the normal value, it indicates hypertriglyceridemia and an increased risk of cardiovascular disease; when it is lower than the normal value, it may be associated with malnutrition or malabsorption.
High-Density Lipoprotein Cholesterol (HDL-C) | Baseline
  Serum level of High-Density Lipoprotein Cholesterol (HDL-C) in mmol/L, which is determined by automatic biochemical analysis. The normal value is ≥1.0 mmol/L. When it is higher than the normal value, it indicates a lower risk of cardiovascular disease; when it is lower than the normal value, it indicates an increased risk of cardiovascular disease.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline
  Serum level of Low-Density Lipoprotein Cholesterol (LDL-C) in mmol/L, which is determined by automatic biochemical analysis. The normal value is <3.4 mmol/L. When it is higher than the normal value, it indicates an increased risk of cardiovascular disease; when it is lower than the normal value, it may be associated with genetic factors or liver dysfunction.
Leptin | Baseline
  Serum level of Leptin in ng/mL, which is determined by automatic biochemical analysis. The normal value is 1.1-27.6 ng/mL. When it is higher than the normal value, it may indicate leptin resistance or obesity; when it is lower than the normal value, it may be associated with malnutrition or low body fat.
Visfatin | Baseline
  Serum level of Visfatin in ng/mL, which is determined by automatic biochemical analysis. The normal value is 10-50 ng/mL. When it is higher than the normal value, it may indicate obesity, insulin resistance, or inflammatory conditions; when it is lower than the normal value, it may be associated with metabolic dysregulation.
Apelin | Baseline
  Serum level of Apelin in pg/mL, which is determined by automatic biochemical analysis. The normal value is 50-200 pg/mL. When it is higher than the normal value, it may indicate cardiovascular stress or metabolic disorders; when it is lower than the normal value, it may be associated with endothelial dysfunction or certain chronic diseases.
Chemerin | Baseline
  Serum level of Chemerin in ng/mL, which is determined by automatic biochemical analysis. The normal value is 50-150 ng/mL. When it is higher than the normal value, it may indicate obesity, insulin resistance, or inflammatory states; when it is lower than the normal value, it may be associated with metabolic dysregulation.
Interleukin-6 (IL-6) | Baseline
  Serum level of Interleukin-6 (IL-6) in pg/mL, which is determined by automatic biochemical analysis. The normal value is <7 pg/mL. When it is higher than the normal value, it indicates an inflammatory response, infection, or autoimmune disease; when it is lower than the normal value, it is generally considered within the normal physiological range.
Interleukin-10 (IL-10) | Baseline
  Serum level of Interleukin-10 (IL-10) in pg/mL, which is determined by automatic biochemical analysis. The normal value is <9.1 pg/mL. When it is higher than the normal value, it may indicate an anti-inflammatory response or certain chronic inflammatory conditions; when it is lower than the normal value, it may be associated with impaired immune regulation.
Transforming Growth Factor-β (TGF-β) | Baseline
  Serum level of Transforming Growth Factor-β (TGF-β) in ng/mL, which is determined by automatic biochemical analysis. The normal value is 5-30 ng/mL. When it is higher than the normal value, it may indicate fibrotic processes, chronic inflammation, or certain cancers; when it is lower than the normal value, it may be associated with impaired tissue repair or immune dysregulation.
Tumor Necrosis Factor-α (TNF-α) | Baseline
  Serum level of Tumor Necrosis Factor-α (TNF-α) in pg/mL, which is determined by automatic biochemical analysis. The normal value is <8.1 pg/mL. When it is higher than the normal value, it indicates systemic inflammation, infection, autoimmune diseases, or certain malignancies; when it is lower than the normal value, it is generally within the normal physiological range.
Irisin | Baseline
  Serum level of Irisin in ng/mL, which is determined by automatic biochemical analysis. The normal value is 3-5 ng/mL. When it is higher than the normal value, it may indicate increased physical activity or improved metabolic status; when it is lower than the normal value, it may be associated with sedentary lifestyle, obesity, or metabolic disorders.
Myostatin | Baseline
  Serum level of Myostatin in ng/mL, which is determined by automatic biochemical analysis. The normal value is 5-15 ng/mL. When it is higher than the normal value, it may indicate muscle wasting conditions or impaired muscle regeneration; when it is lower than the normal value, it may be associated with increased muscle mass or certain metabolic adaptations.
Testosterone | Baseline
  Serum level of Testosterone in ng/dL, which is determined by automatic biochemical analysis. The normal range is 300-1000 ng/dL for adult males and 15-70 ng/dL for adult females. When it is higher than the normal range, it may indicate hyperandrogenism or endocrine disorders; when it is lower than the normal range, it may indicate hypogonadism or age-related decline.
Estrogen | Baseline
  Serum level of Estrogen (Estradiol, E2) in pg/mL, which is determined by automatic biochemical analysis. The normal range varies by gender and life stage: for premenopausal women it is 30-400 pg/mL (varies with menstrual cycle), for postmenopausal women it is <30 pg/mL, and for adult men it is 10-50 pg/mL. When it is higher than the normal range, it may indicate estrogen dominance or certain tumors; when it is lower than the normal range, it may indicate ovarian failure, menopause, or endocrine disorders.
Serum Creatinine | Baseline
  Serum level of Creatinine in μmol/L, which is determined by automatic biochemical analysis. The normal range is 44-133 μmol/L for adult males and 70-106 μmol/L for adult females. When it is higher than the normal range, it may indicate impaired renal function or muscle disorders; when it is lower than the normal range, it may be associated with decreased muscle mass or liver disease.
Cystatin C | Baseline
  Serum level of Cystatin C in mg/L, which is determined by automatic biochemical analysis. The normal range is 0.55-1.02 mg/L. When it is higher than the normal range, it indicates impaired renal function; when it is lower than the normal range, it may be associated with hyperthyroidism or pregnancy.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Hunan, Changsha
  - Suzhou TCM Hospital Affiliated to Nanjing University of Chinese Medicine, Suzhou, Jiangsu
  - Shandong Wendeng Orthopedic Hospital, Weihai, Shandong
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No